CLINICAL TRIAL: NCT03327636
Title: A Prospective Randomized Trial Comparing Ultrasound-guided High Intensity Focused Ultrasound (HIFU) Ablation With Active Surveillance (AS) in the Management of Low-risk Papillary Thyroid Microcarcinoma (PTMC)
Brief Title: A Trial Comparing USG-HIFU vs AS in Management of Low-risk PTMC
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: not start in coming years
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lang Hung Hin, Brian, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 17-175
Record Dates: First submitted 2017-10-25; First posted 2017-10-31 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Papillary Thyroid Microcarcinoma
Keywords: Papillary Thyroid Microcarcinoma; High intensity focused ultrasound; Active surveillance
MeSH Terms: conditions — Papillary Thyroid Microcarcinoma

STUDY DESIGN:
Intervention Model Description: Participants will be arranged into either HIFU group or AS group randomly
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Focused Ultrasound (Experimental): Apply the machine 'Echopulse' with High Intensity Focused Ultrasound to treat the papillary thyroid microcarcinoma.
  Interventions: Device: Echopulse
- Active surveillance (No Intervention): The participants will be monitored by the doctors actively, like more frequent in follow-up to observe their current situation.

INTERVENTIONS:
Device: Echopulse — This is a machine to apply high intensity focused ultrasound to ablation the target zone. In this study, we would apply it to the papillary thyroid microcarcinoma.
  Other Names: High Intensity Focused Ultrasound (HIFU)
  Arms: High Intensity Focused Ultrasound

SUMMARY:
Papillary thyroid microcarcinoma (PTMC) is a common tumor in Hong Kong. Early immediate surgery has traditionally been recommended. However, given its excellent prognosis, some have recommended Active Surveillance (AS) as an alternative. AS involves monitoring the patients who have PTMC until the tumor progresses. On the other hand, a new technology of ablation has been developing to be an alternative treatment for thyroid nodules comparing with traditional surgery, named High intensity focused ultrasound (HIFU). In our previous study, HIFU is proved in shrinking the size of target site by 6 months gradually and effectively.

The investigator hypothesize that HIFU is an effective treatment for PTMC. Compared to AS, HIFU may be a better option as it not only halts disease progression but also has a longer progression-free survival, longer time to tumor progression and is less likely to harbor active disease.

DETAILED DESCRIPTION:
Differentiated thyroid cancer has been rising in incidence and is expected to be a leading cancer by the year 2030 . However, the rise has been mostly attributed to an increased detection of incidentally-discovered papillary thyroid microcarcinoma (PTMC). PTMC is a papillary thyroid carcinoma (PTC) measuring ≤ 10mm in its greatest dimension. Previous screening and autopsy studies have confirmed these lesions are common and could be found in up to 15% of normal healthy individuals.

However, since the incidence of clinically-significant PTC has historically been <0.5% (i.e. 100 times less than the occult rate), most occult PTMCs probably do not cause harm in one's life-time and could be safely observed without immediate surgery.

As a result, several groups of investigators worldwide began evaluating the feasibility and safety of observing PTMC without surgery. Rather than offering immediate surgery, well selected patients with low-risk PTMC (i.e. no extrathyroidal extension, nodal and distant metastases) were followed with regular ultrasound (USG) alone and only proceeded to definitive to surgery when the PTMC showed progression. As expected, >90% PTMCs did not progress and of those who progressed and had surgery, all were cured. This meant even when the initial surgery was deferred, there was no compromise in the chance of cure.

With a recent shift towards a more conservative approach in the management of PTC, it has become increasingly accepted that perhaps active surveillance (AS) might be a safe alternative in well selected low-risk PTMCs.

However, despite the fact that AS is a viable alternative, there are issues and challenges. First, although the majority of occult tumors do not progress initially, the accumulative risk of tumor progression increases with time. From an analysis of the 1479 PTMCs observed over 5 years, 212 (14.3%) eventually met the progression criteria (such as tumor enlargement, local invasion, new lymph node metastasis or becoming clinical disease) and had surgery. Therefore, with longer observation, a greater proportion of patients would end up having surgery. Second some patients tend to find it difficult to accept AS as a treatment. Even if they do initially, the "wait and see" approach may distress patients leading to non-compliance. To date, little is known how this may affect patients' well-being and health-related quality of life (HRQOL) over time. Third, since there are no clinical or molecular parameters to predict which tumors are more likely to progress, patients often need life-long follow-up. However, this may be challenging because patients may move to different places. Lastly, there are now less invasive, non-surgical options available to potentially eradicate PTMCs. Image-guided thermal ablation (IGTA) using laser ablation or radiofrequency ablation appears promising. With technological advances, they may eventually replace surgery in the future. However, reports have so far been non-randomized, uncontrolled and short follow-up. Furthermore, despite being less-invasive, they still require a small skin incision.

High intensity focused ultrasound (HIFU) is a form of IGTA that needs no skin incision or needle insertion and so, is a truly noninvasive treatment. Under USG guidance, it is able to cause irreversible tissue destruction deep to the skin and subcutaneous layer. Apart from being non-invasive, it is less dependent on the operator's skill as the treatment could be controlled by an automated program. In fact, HIFU is highly successful in a number of solid cancers. In the thyroid, it induces tissue damage via the cavitation and thermal effects. To date, several groups (including us) have confirmed that HIFU ablation is highly effective in inducing shrinkage of benign thyroid nodules.

ELIGIBILITY:
Inclusion Criteria:

* Have a thyroid nodule ≤10mm in the largest dimension that is confirmed on FNAC to be PTC (Bethesda class VI cytology) or suspicious of PTC (Bethesda V cytology). For the latter, the nodule needs to have an additional suspicious sonographic feature (i.e. marked hypoechogenicity, irregular margins, height-to-wide ratio >1 and intravascular microcalcifications);
* Have not expressed a strong desire for immediate surgery after PTMC has been confirmed.

Exclusion Criteria:

* Age ≤ 18 or ≥ 75 years old;
* Have another thyroid nodule that is either indeterminate or malignant on FNAC;
* Have concomitant hypo- or hyperthyroidism (i.e. thyroid stimulating hormone (TSH) and/or free thyroxine levels outside the normal ranges)
* Have sonographic evidence of chronic lymphocytic thyroiditis (because this generally makes it difficult to assess and reassess tumor size accurately on USG alone)
* Have a tumor considered not suitable for AS. This includes a PTMC with extrathyroidal extension, concomitant nodal or distant metastasis or a PTMC located within 3mm from trachea-esophageal groove or recurrent laryngeal nerve.
* Have a condition considered not suitable for HIFU treatment (pregnancy, history of neck irradiation, known contralateral vocal cord palsy, a tumor with coarse, macroscopic intranodular calcifications or located outside the treatable depth of 5-30 mm from the skin, family history of non-medullary thyroid carcinoma and medical conditions precluding intravenous sedation).

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of tumors exhibiting disease progression | 24 months
  To compare the proportion of patients with PTMC exhibiting signs of progression between HIFU and AS group at 24 months

SECONDARY OUTCOMES:
Median duration of progression-free survival | 24 months
  To examine the median duration of progression-free survival within 2 years
Change in tumor volume | 24 months
  Tumor volume change from baseline (%) at 2 years
Proportion of patients with active disease | 24 months
  The proportion of patients with active disease confirmed by re-biopsy and CEUSG (%) at 2 years
Proportion of patients undergoing planned and unplanned thyroidectomy | 24 months
  To calculate the proportion of patients who undergoing thyroidectomy in planned or unplanned.
Health related quality of life (HRQOL) | 24 months
  To examine participants HRQOL during the study with a questionnaire combined with different measurement tools: SF-12 (12-Item Short Form Health Survey), SF-6D (Short Form 6 Dimensions), EQ-5D-5L (EuroQoL 5 Dimensions 5 Levels) and FACT-G (Functional Assessment of Cancer Therapy - general scale). The total score would be the health score of participants, as high score as high quality of life.
Incidence of potential side-effects from intensity focused ultrasound treatment | 24 months
  To examine any treatment-related side-effects after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hung Hin, Brian Lang, MBBS (Hons), Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Background] Davies L, Welch HG. Increasing incidence of thyroid cancer in the United States, 1973-2002. JAMA. 2006 May 10;295(18):2164-7. doi: 10.1001/jama.295.18.2164. PMID 16684987
- [Background] Vaccarella S, Franceschi S, Bray F, Wild CP, Plummer M, Dal Maso L. Worldwide Thyroid-Cancer Epidemic? The Increasing Impact of Overdiagnosis. N Engl J Med. 2016 Aug 18;375(7):614-7. doi: 10.1056/NEJMp1604412. No abstract available. PMID 27532827
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Ito Y, Miyauchi A, Kihara M, Higashiyama T, Kobayashi K, Miya A. Patient age is significantly related to the progression of papillary microcarcinoma of the thyroid under observation. Thyroid. 2014 Jan;24(1):27-34. doi: 10.1089/thy.2013.0367. Epub 2013 Nov 14. PMID 24001104
- [Background] Sugitani I, Toda K, Yamada K, Yamamoto N, Ikenaga M, Fujimoto Y. Three distinctly different kinds of papillary thyroid microcarcinoma should be recognized: our treatment strategies and outcomes. World J Surg. 2010 Jun;34(6):1222-31. doi: 10.1007/s00268-009-0359-x. PMID 20066418
- [Background] Ito Y, Miyauchi A, Inoue H, Fukushima M, Kihara M, Higashiyama T, Tomoda C, Takamura Y, Kobayashi K, Miya A. An observational trial for papillary thyroid microcarcinoma in Japanese patients. World J Surg. 2010 Jan;34(1):28-35. doi: 10.1007/s00268-009-0303-0. PMID 20020290
- [Background] Lang BH, Wong CK. A cost-effectiveness comparison between early surgery and non-surgical approach for incidental papillary thyroid microcarcinoma. Eur J Endocrinol. 2015 Sep;173(3):367-75. doi: 10.1530/EJE-15-0454. Epub 2015 Jun 23. PMID 26104754
- [Background] National Cancer Comprehensive Network (NCCN Guidelines) 2015 Thyroid carcinoma. Version 2. 2015. Available: http://www.nccn.org/professionals/physician_gls/f_guidelines.asp [Accessed on 16th February 2016]
- [Background] Perros P, Boelaert K, Colley S, Evans C, Evans RM, Gerrard Ba G, Gilbert J, Harrison B, Johnson SJ, Giles TE, Moss L, Lewington V, Newbold K, Taylor J, Thakker RV, Watkinson J, Williams GR; British Thyroid Association. Guidelines for the management of thyroid cancer. Clin Endocrinol (Oxf). 2014 Jul;81 Suppl 1:1-122. doi: 10.1111/cen.12515. No abstract available. PMID 24989897
- [Background] Brito JP, Ito Y, Miyauchi A, Tuttle RM. A Clinical Framework to Facilitate Risk Stratification When Considering an Active Surveillance Alternative to Immediate Biopsy and Surgery in Papillary Microcarcinoma. Thyroid. 2016 Jan;26(1):144-9. doi: 10.1089/thy.2015.0178. Epub 2015 Nov 5. PMID 26414743
- [Background] Papini E, Guglielmi R, Gharib H, Misischi I, Graziano F, Chianelli M, Crescenzi A, Bianchini A, Valle D, Bizzarri G. Ultrasound-guided laser ablation of incidental papillary thyroid microcarcinoma: a potential therapeutic approach in patients at surgical risk. Thyroid. 2011 Aug;21(8):917-20. doi: 10.1089/thy.2010.0447. Epub 2011 May 19. PMID 21595556
- [Background] Zhang M, Luo Y, Zhang Y, Tang J. Efficacy and Safety of Ultrasound-Guided Radiofrequency Ablation for Treating Low-Risk Papillary Thyroid Microcarcinoma: A Prospective Study. Thyroid. 2016 Nov;26(11):1581-1587. doi: 10.1089/thy.2015.0471. Epub 2016 Aug 18. PMID 27445090
- [Background] Monchik JM, Donatini G, Iannuccilli J, Dupuy DE. Radiofrequency ablation and percutaneous ethanol injection treatment for recurrent local and distant well-differentiated thyroid carcinoma. Ann Surg. 2006 Aug;244(2):296-304. doi: 10.1097/01.sla.0000217685.85467.2d. PMID 16858194
- [Background] She WH, Cheung TT, Jenkins CR, Irwin MG. Clinical applications of high-intensity focused ultrasound. Hong Kong Med J. 2016 Aug;22(4):382-92. doi: 10.12809/hkmj154755. Epub 2016 Jul 6. PMID 27380753
- [Background] Esnault O, Franc B, Chapelon JY. Localized ablation of thyroid tissue by high-intensity focused ultrasound: improvement of noninvasive tissue necrosis methods. Thyroid. 2009 Oct;19(10):1085-91. doi: 10.1089/thy.2009.0121. PMID 19803790